CLINICAL TRIAL: NCT05491512
Title: Major Radiation Dose De-Escalation Concurrent With Chemotherapy for Human Papilloma Virus Associated Oropharyngeal Carcinoma
Brief Title: A Study of Reduced Radiation Therapy and Standard-of-Care Chemotherapy in People With HPV-Positive Throat Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-215
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: HPV; Throat Cancer; Oropharyngeal Carcinoma; Oropharyngeal Cancer; Human Papilloma Virus
Keywords: HPV-Positive Throat Cancer; HPV; Throat Cancer; Human Papilloma Virus; Oropharyngeal Carcinoma; Oropharyngeal Cancer; Radiation Therapy; 22-215; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Radiation; Cisplatin; Carboplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A (Experimental): Participants diagnosed with hypoxia negative human papilloma virus (HPV) associated oropharyngeal carcinoma (OPC)
  Interventions: Diagnostic Test: 18 F-FMISO PET/CT; Radiation: Radiation; Drug: Cisplatin; Drug: Carboplatin; Drug: 5-fluorouracil
- Cohort B (Experimental): Participants diagnosed with hypoxia negative human papilloma virus (HPV) associated oropharyngeal carcinoma (OPC). Participants in Cohort B will receive 1 cycle of carboplatin and Paclitaxol the same week of the start of radiation. Paclitaxel can be substituted with Abraxane (Albumin-bound Paclitaxel). Paclitaxel can be substituted with Abraxane and the dose will be 50mg/m^2. For Cohort B, patients over 70yrs will be able to enroll regardless of Cisplatin or carboplatin/5-fluorouracil (FU) eligibility.
  Interventions: Diagnostic Test: 18 F-FMISO PET/CT; Radiation: Radiation; Drug: Cisplatin; Drug: Carboplatin; Drug: 5-fluorouracil
- Cohort C (Experimental): Participants diagnosed with hypoxia negative human papilloma virus (HPV) associated oropharyngeal carcinoma (OPC). For participants in Cohort C where induction chemotherapy is used, additional pre-treatment 18F-FMISO PET and post induction pre radiation FMISO PET Scans will be obtained. These patients will start with induction chemotherapy of carboplatin, paclitaxel with or without cetuximab for 6 weeks and follow the same precision chemoradiation algorithm as Cohort A. A window of +/- 2 days is acceptable during the induction phase Paclitaxel can be substituted with Abraxane (Albumin-bound Paclitaxel). For patients who cannot tolerate paclitaxel, Abraxane and the dose will be at 100mg/m^2.
  Interventions: Diagnostic Test: 18 F-FMISO PET/CT; Radiation: Radiation; Drug: Cisplatin; Drug: Carboplatin; Drug: 5-fluorouracil
- Cohort D (Experimental): Participants diagnosed with hypoxia negative human papilloma virus (HPV) associated oropharyngeal carcinoma (OPC). Cohort D will just have T1- T2N0 participants. Paclitaxel can be substituted with Abraxane (Albumin-bound Paclitaxel). Will follow the guidelines for Cohort A and Cohort B for chemotherapy options.
  Interventions: Diagnostic Test: 18 F-FMISO PET/CT; Radiation: Radiation; Drug: Cisplatin; Drug: Carboplatin; Drug: 5-fluorouracil

INTERVENTIONS:
Diagnostic Test: 18 F-FMISO PET/CT — The 18F-FMISO PET/CT Scan Protocol consists first of an IV bolus injection of approximately 5-10 mCi of the radiotracer. At between 150-180 mins post injection, 18F-FMISO images will be acquired.
Radiation: Radiation — Total Radiation Dose (over 3 weeks) 30Gy** in 2 Gy per fraction
Drug: Cisplatin — Concurrent chemotherapy (2 cycles) will be given. At the start of week 1 of radiation, subjects will receive cisplatin 100 mg/m2 intravenously. They may be given for 2 consecutive days (50 mg/m2 each day for a total dose 100 mg/m2 ), typically on days 1 and 2, or as a single dose, typically on day 1.
Drug: Carboplatin — If cisplatin cannot be given at 100 mg/m2 for either cycle 1 or cycle 2, the investigator may use a regimen with carboplatin and 5-Fluorouracil in its place. Carboplatin will be given at a dose of AUC 1.25 intravenously daily x 4 days starting on day 1 of the cycle (total dose of AUC 5). 5-Fluorouracil will be given at a dose of 600 mg/m2 intravenous infusion over 24 hours daily x 4 days (total dose of 2400 mg/m2 intravenous infusion over 96 hours).
  (Cohort B to start carboplatin (AUC 1.5) and paclitaxel 45 mg/m2 at the start of RT)
Drug: 5-fluorouracil — If cisplatin cannot be given at 100 mg/m2 for either cycle 1 or cycle 2, the investigator may use a regimen with carboplatin and 5-Fluorouracil in its place. Carboplatin will be given at a dose of AUC 1.25 intravenously daily x 4 days starting on day 1 of the cycle (total dose of AUC 5). 5-Fluorouracil will be given at a dose of 600 mg/m2 intravenous infusion over 24 hours daily x 4 days (total dose of 2400 mg/m2 intravenous infusion over 96 hours).

SUMMARY:
The purpose of this study is to find out if lower doses of radiation may help reduce the side effects of radiation therapy in combination with standard-of-care chemotherapy in people with HPV-positive throat cancer. The chemotherapy drugs used in this study include cisplatin, carboplatin, and 5-fluorouracil (5- FU), paclitaxel and abraxane- (Albumin-bound Paclitaxel).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of HPV associated squamous cell carcinoma of the oropharynx (tonsil, base of tongue, or oropharyngeal walls) from biopsy, surgical resection or excisional biopsy regardless of margin status.

  1. Squamous cell carcinoma of the neck of unknown primary is allowed with excision biopsy of a lymph node (or core biopsy) or consent from the PI or co-PI
  2. Patient must have excisional biopsy or core biopsy done in order to be on protocol
* Subjects must have clinically or radiographically evident measurable gross disease at either the primary tumor site or nodal stations.
* Oropharyngeal Carcinoma (AJCC, 7th ed.) without evidence of distant metastasis based on FDG PET/CT.
* CT or MRI of the neck with and without contrast Note: A CT scan of neck and/or a PET/CT performed for the purposes of radiation planning may serve as planning tools.
* ECOG Performance Status of 0-2 or KPS ≥ 50
* Age ≥ 18 Patients over 70yrs will be able to enroll in Cohort B only).
* Adequate hematologic function within 30 days prior to registration, defined as follows:

  1. White Blood Count (WBC) ≥ 2 K/mcL
  2. Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3
  3. Platelets ≥ 100,000 cells/mm3
  4. Hemoglobin ≥ 8.0 g/dl; Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable
* Adequate renal function within 30 days prior to registration, defined as follows:

  1. Serum creatinine < 1.5 mg/dl or creatinine clearance (CC) ≥ 50 ml/min determined by 24-hour collection or estimated by Cockcroft-Gault formula: CCr male = [(140 - age) x (wt in kg)] [(Serum Cr mg/dl) x (72)] CCr female = 0.85 x (CrCl male)

Note: Patients who cannot tolerate cisplatin or carboplatin/5FU based on clinical judgment will receive carboplatin and paclitaxel Paclitaxel can be substituted with Abraxane (Albumin-bound Paclitaxel).

* Adequate hepatic function within 30 days prior to registration, defined as follows:

  1. Bilirubin < 2 mg/dl
  2. AST or ALT < 3 x the upper limit of normal

Note: Exceptions can be made with PI and/or Co-Pi approval for patients to enroll on trial with a higher Bilirubin level such as Gilbert's Syndrome.

Note: Patients who cannot tolerate cisplatin or carboplatin/5FU based on clinical judgment will receive carboplatin and paclitaxel. Paclitaxel can be substituted with Abraxane (Albumin-bound Paclitaxel).

* Negative serum pregnancy test within 14 days prior to registration for women of childbearing potential
* The subject must provide study-specific informed consent prior to study entry
* Subject able to undergo MRI scans except for major medical contraindications like presence of a pacemaker or approved by the PI or the CO-PI that the subject does not need to undergo MRI scans

Exclusion Criteria:

* Subjects with prior head and neck radiation therapy
* Subjects with simultaneous primary cancers outside of the oropharynx

  a. Note: Exceptions can be made for patients with simultaneous primaries outside the oropharynx if determined by the PI/Co-PI the patient can proceed with protocol activities.
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for 3 years or if cure rate from treatment at 5 years to be 90% or greater
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable
* Severe, active co-morbidity defined as follows: (exceptions can be made if approved by the PI and/or co-PI)

  1. Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  2. Transmural myocardial infarction within the last 6 months
  3. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  4. Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration
  5. Hepatic Insufficiency resulting in clinical jaundice and/or coagulation defects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2026-08-04 (Estimated); Study Completion 2026-08-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with any locoregional recurrences | 2 years
  The primary objective of this protocol is to demonstrate that the 2 year locoregional control for these subjects treated with a major de-escalated radiation dose of 30Gy is acceptable as compared to historical locoregional control rate for subjects treated with the current standard chemoradiation at 70Gy. To examine if subjects receiving 30Gy have an acceptable treatment outcome when compared to the radiation of 70Gy both in the setting of concurrent chemotherapy, we will test the hypothesis that H0: P<=85% vs H1: P>85%, where P represents the 2-year locoregional control rate.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lee, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Cancer Center at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center at Suffolk-Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org